CLINICAL TRIAL: NCT02278055
Title: Phase II Open, Non-Randomized Trial Assessing Pain Efficacy With Radium-223 in Symptomatic Metastatic Castration-Resistant Prostate Cancer
Brief Title: Non-Randomized Trial Assessing Pain Efficacy With Radium-223 in Symptomatic Metastatic Castration-Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: University of North Carolina (Other); New York Presbyterian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-098; c13-124 (Other: Prostate Cancer Clinical Trials Consortium)
Record Dates: First submitted 2014-10-25; First posted 2014-10-29 (Estimated); Results first posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2021-08

CONDITIONS: Metastatic Prostate Cancer; Pain
Keywords: Radium-223; 14-098; Prostate Cancer Clinical Trials Consortium
MeSH Terms: conditions — Prostatic Neoplasms; Pain | interventions — Radium-223

ARMS (1):
- Radium-223 (Experimental): Radium Ra 223 dichloride will be administered as a bolus intravenous (IV) injection (up to 1 minute) at intervals of every 4 weeks for up to 6 cycles. The dosage of Radium Ra 223 dichloride after implementation of the new 2015 NIST standard is 55kBq/kg body weight.
  Interventions: Drug: Radium-223

INTERVENTIONS:
Drug: Radium-223

SUMMARY:
The purpose of this study is to find out if Radium-223 is effective in reducing cancer pain within 12 weeks of treatment. In order to see if Radium-223 is effective, the patient's level of pain will be followed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 18 years of age and above
* Histological or cytological proof of prostate adenocarcinoma
* Castrate serum testosterone level: ≤50 ng/dL (≤1.7 nmol/L)
* Patients who have experienced disease progression despite initial hormonal therapy, either by orchiectomy or by using a GnRH agonist in combination with an anti-androgen, must first progress through anti- androgen withdrawal prior to being eligible. The minimum time frame to document failure of anti-androgen withdrawal will be four weeks. Patients on second-line (or beyond) hormonal maneuvers, and patients who had no PSA decline on combined androgen blockade as first line therapy, need not progress through AAW in order to be eligible.
* Known progressive castration-resistant disease, defined as:

  * Serum PSA progression defined as two consecutive increases in PSA over a previous reference value within 6 months of first treatment, each measurement at least one week apart. Serum PSA at screening ≥ 2 ng/mL or
  * Documented appearance of new lesions by bone scintigraphy
* ECOG Performance Status of 0-2 2 or more bone metastases demonstrated on bone scintigraphy
* Pain at baseline as measured by a BPI worst pain score average of ≥ 3. The BPI worst pain score average will be based on the worst pain scores completed by the patient in the 7 consecutive pretreatment days. A minimum of 4 days of pain scores must be completed by the patient in the 7 day window in order to calculate the average worst pain score. The investigator will optimize the subject's pain regimen prior to study entry.
* Normal organ function with acceptable initial laboratory values:

  * WBC ≥ 3 x 109 /L
  * ANC ≥ 1.5 x 109 /L
  * Platelets ≥ 100 x 109 /L
  * Hemoglobin ≥ 9.0 g/dL
  * Creatinine < 1.5 x institutional upper limit of normal (ULN)
  * Bilirubin ≤ 1.5 x ULN
  * AST/ALT ≤ 2.5 x ULN
  * Albumin > 25 g/L
* All acute toxicities as a result of any prior treatment must have resolved to NCI-CTCAE v4.0 Grade 1 or less at the time of signing the Informed Consent Form (ICF) [Note: Ongoing grade 2 neuropathy as a result of treatment with a cytotoxic chemotherapy regimen is permitted]
* Life expectancy of at least 6 months
* Willing and able to provide written informed consent and HIPAA authorization for the release of personal health information NOTE: HIPAA authorization may be either included in the informed consent or obtained separately
* Willing and able to comply with the protocol, including follow-up visits, examinations as well as having the ability to self-report pain and fatigue using a Patient Reported Outcome (PRO) instrument
* Willingness to use adequate methods of contraception beginning at the signing of the ICF until at least 30 days after the last dose of study drug

Exclusion Criteria:

* Prior exposure to Radium-223
* Received an investigational therapy within the 4 weeks prior to registration or is scheduled to receive one during the treatment period
* Received a new anti-cancer agent within 4 weeks prior to registration
* Received external beam radiotherapy within 4 weeks prior registration
* Received systemic therapy with radionuclides (e.g. strontium-89, samarium-153, rhenium-186 or rhenium-188) for the treatment of bone metastases
* Treatment with cytotoxic chemotherapy within 4 weeks prior to registration
* Symptomatic nodal disease, i.e. scrotal, penile or leg edema. Visceral metastases (including cerebral metastases) from CRPC (>2 lung and/or liver metastases [size ≥2cm]; Lymphadenopathy exceeding 6 cm in short-axis diameter or any size pelvic lymphadenopathy if it is thought to be a contributor to concurrent hydronephrosis), as assessed by CT, MRI or chest X-ray within the 8 weeks prior registration.
* Concurrent chemotherapy. Patients may be on other non-chemotherapy anti-cancer treatments, per FDA labeling of Radium-223, provided that these are not changed during the primary pain assessment period Major surgery within 30 days prior to registration.
* Imminent spinal cord compression based on clinical findings and/or magnetic resonance imaging (MRI). Treatment should be completed for spinal cord compression.
* Patients with a, "currently active," second malignancy other than non-melanoma skin cancers or non-invasive bladder cancers or other in-situ or non-invasive malignancies. Patients who have completed therapy for a prior malignancy and are free of disease for ≥3 years are eligible.
* Any other serious illness or medical condition, such as but not limited to:

  * Any infection ≥ National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 4.03 Grade 2
  * Cardiac failure New York Heart Association (NYHA) III or IV
  * Crohn's disease or ulcerative colitis
  * Bone marrow dysplasia
  * Fecal incontinence
* Any other condition which, in the opinion of the Investigator, would make the subject unsuitable for trial participation
* NOTE: Any patient found to be ineligible prior to treatment initiation will require re-screening.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2014-10-08 (Actual); Primary Completion 2022-02-02 (Actual); Study Completion 2022-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Morris, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital-Weill Medical College of Cornell University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Radium-223: Radium Ra 223 dichloride will be administered as a bolus intravenous (IV) injection (up to 1 minute) at intervals of every 4 weeks for up to 6 cycles. The dosage of Radium Ra 223 dichloride after implementation of the new 2015 NIST standard is 55kBq/kg body weight.
  Radium-223
Period: Overall Study
Arm/Group | Radium-223
Started | 29
Completed | 21
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 4

BASELINE CHARACTERISTICS:
Arm/Group | Radium-223
Number analyzed (Participants) | 29
Age, Continuous [Median (Full Range); unit: years] | 69 [52 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With 30% Decline in the Brief Pain Inventory (BPI) Worst Pain Item From Baseline to Week 8
Description: Defined as a 30% decline in the Brief Pain Inventory/BPI worse pain item from baseline to week 8, with a confirmed reduction at week 12 without an escalation of the subject's pain regimen from Step 1 to Step 2 or Step 2 to Step 3 of the WHO analgesic ladder.) The baseline BPI worst pain score average will be based on the worst pain scores completed by the participant in the 7 consecutive pretreatment days. A minimum of 4 days of pain scores must be completed by the participant in the 7 day window in order to calculate the average worst pain score. The BPI scale defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain.
Time Frame: 8 weeks
Measure: Number; unit: Percentage of pts w/pain improvement
Arm/Group | Radium-223
Number analyzed (Participants) | 21
Percentage of pts w/pain improvement | 11

2. Secondary Outcome: Number of Participants With Changes in Bone Alkaline Phosphatase (ALP)
Description: Number of participants with changes from baseline to 12 weeks (or earlier for those who discontinue study therapy). Maximum change (rise or fall) in bone Alkaline phosphatase (ALP) during the treatment period reported.
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 29
Participants
  Count of non pain responders with consecutive decrease in Bone Alkaline Phosphatase | 18
  Count of pain responders with consecutive decrease in Bone Alkaline Phosphatase | 9
  Count of participants with no change | 2

3. Secondary Outcome: Number of Participants With Changes in Other Bone Markers:
Description: Serum C-telopeptide (sCTX-1) N-terminal propeptide of procollagen type 1 (PINP) Changes in total-ALP will be defined as for bone-ALP above
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Radium-223
Number analyzed (Participants) | 29
Participants
  Count of pain responder participants with consecutive decrease in N-terminal propeptide | 9
  Count of participants with no consecutive decrease in N-terminal propeptide | 20

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Radium-223
All-Cause Mortality (participants affected / at risk) | 5/29
Serious Adverse Events (participants affected / at risk) | 11/29
Other Adverse Events (participants affected / at risk) | 22/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radium-223 (N=29)
Diarrhea (Gastrointestinal disorders) | 1
Esophageal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Malaise (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Fracture (Injury, poisoning and procedural complications) | 1
Weight loss (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 2
Buttock pain (Musculoskeletal and connective tissue disorders) | 1
Neoplasms ben/mal/unk (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Radiculitis (Nervous system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Radium-223 (N=29)
Anemia (Blood and lymphatic system disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hypoalbuminemia (Metabolism and nutrition disorders) | 5
Alkaline phosphatase increased (Investigations) | 3
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3
White blood cell decreased (Investigations) | 3
Creatinine increased (Investigations) | 2
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 2
INR increased (Investigations) | 2
Platelet count decreased (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-01): https://cdn.clinicaltrials.gov/large-docs/55/NCT02278055/Prot_SAP_000.pdf